CLINICAL TRIAL: NCT01271907
Title: Phase II Study of Metastatic Melanoma Using a Nonmyeloablative Lymphodepleting Regimen Followed by Melanoma-Reactive T-Cells Sensitized in Vitro With Peptide-Pulsed Drosophila Cells
Brief Title: Drosophila-generated CTL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to withdrawal of CRADA partner.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Yang, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110052; 11-C-0052
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Cutaneous Melanoma
Keywords: Skin Cancer; Malignancy; Immunotherapy; Melanoma Peptides; Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Neoplasms | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 0 (Experimental): Drosophila generated CTL + SQ IL-2 Drug: 1 fludarabine, cyclophosphamide, Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ peripheral blood lymphocytes (PBL) (CTL-05), aldesleukin Fludarabine 25 mg/m^2 x 5 days Cyclophosphamide 60 mg/kg intravenous (IV) x2 days, Up to 1x10e10 CTL-05 cells Aldesleukin 125,000 IU/kg/dose as a daily subcutaneous injection
  Interventions: Drug: fludarabine; Drug: cyclophosphamide; Drug: Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ PBL; Drug: Aldesleukin
- Cohort 1 (Experimental): 2 Experimental Lymphodepleting regimen +Cells+Low dose IL-2 Drug: 2 fludarabine, cyclophosphamide, Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ peripheral blood lymphocytes (PBL), aldesleukin Fludarabine 25 mg/m^2 x 5 days Cyclophosphamide 60 mg/kg intravenous (IV) x2 days, Up to 1x10e10 CTL-05 cells Aldesleukin 125,000 IU/kg/dose as a daily subcutaneous injection
  Interventions: Drug: fludarabine; Drug: cyclophosphamide; Drug: Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ PBL; Drug: Aldesleukin
- Cohort 2 (Experimental): 1 Experimental Lymphodepleting regimen +Cells Drug: 3 fludarabine, cyclophosphamide, Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ peripheral blood lymphocytes (PBL) Fludarabine 25 mg/m^2 x 5 days Cyclophosphamide 60 mg/kg intravenous (IV) x2 days, Up to 1x10e10 CTL-05 cells
  Interventions: Drug: fludarabine; Drug: cyclophosphamide; Drug: Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ PBL; Drug: Aldesleukin

INTERVENTIONS:
Drug: fludarabine — Fludarabine 25 mg/m^2 x 5 days
  Other Names: Fludara
Drug: cyclophosphamide — Cyclophosphamide 60 mg/kg intravenous (IV) x 2 days
  Other Names: Cytoxan
Drug: Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ PBL — Up to 1x10e10 CTL-05 cells
Drug: Aldesleukin — Aldesleukin 125,000 IU/kg/dose as a daily subcutaneous injection
  Other Names: IL-2

SUMMARY:
Background:

* Recent cancer treatment studies have shown that altering a cancer patient's own white blood cells may help the immune system fight the cancer. In all of these studies, participants donate their own white blood cells through a procedure called leukapheresis, and the cells are altered in the laboratory and given back to the participants. After the cells are given, the patients receive aldesleukin (IL-2) to help the tumor fighting cells stay alive longer. For individuals with metastatic melanoma, pieces of melanoma proteins may be added to the collected white blood cells to help the immune system recognize and attack the cancer cells.
* Researchers are interested in testing a new process in which cells from fruit flies (Drosophila) are used to help the melanoma proteins attach to the white blood cells. The fruit fly cells die off shortly after the proteins are introduced to the white blood cells. Researchers are also interested in determining whether IL-2 treatment is necessary after this new cancer treatment process.

Objectives:

* To test the safety and effectiveness of modified white blood cells (Drosophila-generated CTL) as a treatment for metastatic melanoma that has not responded to standard treatments.
* To determine whether IL-2 treatment improves the effectiveness of Drosophila-generated cytolytic T lymphocytes (CTL).

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with metastatic melanoma that has not responded to previous IL-2 treatment.

Design:

* Participants will be screened with a physical examination and medical history, tumor imaging studies, and heart and lung function tests.
* Prior to treatment, participants will have an intravenous catheter inserted into the chest to administer the study drugs.
* Participants will have leukapheresis to provide white blood cells for laboratory modification.
* Seven days before the start of the treatment, participants will be admitted to the hospital to have chemotherapy with cyclophosphamide and fludarabine. These drugs will suppress the immune system to improve the effects of the treatment.
* One to four days after the last dose of chemotherapy, participants will receive the modified cells. Participants in the group that will receive IL-2 will begin to receive the treatment 24 hours after the cell infusion, every day for 5 days. All participants will receive filgrastim injections to help the body produce more white blood cells.
* Participants will recover in the hospital for about 7 to 12 days after the cell infusion or the last dose of IL-2. Participants will continue to receive medications and provide blood and tumor samples for testing.
* Participants will have regular followup visits to assess the effects of the treatment.

DETAILED DESCRIPTION:
Background:

* Adoptive transfer studies in patients with metastatic melanoma following lymphodepletion have resulted in up to 50% objective response rates with a 10-15% rate of complete responses.
* A novel method involves the use of insect cell lines which do not express any native major histocompatibility complex (MHC) molecules.
* When stably transfected with human MHC molecules and appropriate adhesion and costimulatory molecules, a Drosophila cell line can potently stimulate tumor-reactivity in vitro from human peripheral blood lymphocytes (PBL).
* The current proposed transfer of Drosophila-cell stimulated autologous cluster of differentiation 8 (CD8) plus PBL administered in conjunction with a lymphodepleting preparative regimen, with or without low-dose aldesleukin would represent a significantly novel approach to adoptive immunotherapy.

Objectives:

* To determine whether infusion of CD8+ autologous PBL sensitized in vitro with peptide pulsed HLA-A2-expressing Drosophila cells (CTL-05) and administered in combination with a lymphodepleting preparative regimen and supportive systemic aldesleukin can result in clinical tumor regression in human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2+) patients with metastatic melanoma.
* To determine the safety of the above regimen.
* To investigate the contribution of low-dose systemic aldesleukin to cell efficacy.

Eligibility:

Patients who are HLA-A*0201 positive and 18 years of age or older must have

* metastatic melanoma with measurable disease
* been previously treated with aldesleukin for melanoma;
* normal basic laboratory values.

Patients may not have:

* concurrent major medical illnesses;
* any form of primary or secondary immunodeficiency;
* requirement for systemic steroid therapy

Design:

* The first 20 patients enrolled (cohort 0) will receive a non-myeloablative lymphocyte depleting preparative regimen followed by administration of intravenous CTL-05 and low-dose subcutaneous aldesleukin (daily for 5 days).
* If 3 or more of the 20 patients respond, subsequent patients will be randomized between two cohorts. Patients in cohort 1 will receive a non-myeloablative lymphocyte depleting preparative regimen followed by administration of CTL-05 and low-dose subcutaneous aldesleukin (daily for 5 days). Patients in Cohort 2 will receive a non-myeloablative lymphocyte depleting preparative regimen followed by administration of CTL-05 and NO subsequent aldesleukin.
* A complete evaluation will be conducted 8 weeks (plus or minus 2 weeks) after the initiation of chemotherapy. The trial will be conducted using a small Simon MinMax Phase II design in the initial phase and a Simon optimal design in the second phase. A maximum of 35 patients may be accrued to each of cohorts 1 and 2. If no responses are seen in the first 13 patients receiving no systemic aldesleukin, then accrual to that cohort will cease. Total enrollment may be up to 90 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic cutaneous melanoma with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
  2. Previously received high dose-aldesleukin and have been either non-responders (progressive disease) or have recurred.
  3. Patients with 3 or less brain metastases are eligible. Note: If lesions are symptomatic or greater than or equal to 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible.
  4. Greater than or equal to 18 years of age.
  5. Able to understand and sign the Informed Consent Document
  6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  7. Life expectancy of greater than three months.
  8. Patients of both genders must be willing to practice a highly effective method of birth control during and for four months following treatment
  9. Patients must be HLA-A*0201 positive
  10. Serology:

      1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
      2. Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
  11. Hematology:

      1. Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
      2. White blood cell (WBC) (> 3000/mm^3).
      3. Platelet count greater than 100,000/mm^3.
      4. Hemoglobin greater than 8.0 g/dl.
  12. Chemistry:

      1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  13. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for hypothyroidism, alopecia, or vitiligo).
  14. Six weeks must have elapsed since prior anti-CTLA4 antibody therapy to allow antibody levels to decline.
  15. Patients who have previously received anti-CTLA4 antibody must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Active systemic infections, coagulation disorders or other active major medical illnesses.
2. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
3. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
4. Requirement for systemic steroid therapy
5. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
6. History of coronary revascularization or ischemic symptoms
7. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
8. Documented LVEF of less than or equal to 45% tested in patients with:

   1. Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   2. Age greater than or equal to 60 years old
9. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

   1. A prolonged history of cigarette smoking (20 pk/yrs of smoking)
   2. Symptoms of respiratory dysfunction
10. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04-15 (Actual); Primary Completion 2011-12-08 (Actual); Study Completion 2011-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Yang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balch CM, Soong SJ, Gershenwald JE, Thompson JF, Reintgen DS, Cascinelli N, Urist M, McMasters KM, Ross MI, Kirkwood JM, Atkins MB, Thompson JA, Coit DG, Byrd D, Desmond R, Zhang Y, Liu PY, Lyman GH, Morabito A. Prognostic factors analysis of 17,600 melanoma patients: validation of the American Joint Committee on Cancer melanoma staging system. J Clin Oncol. 2001 Aug 15;19(16):3622-34. doi: 10.1200/JCO.2001.19.16.3622. PMID 11504744
- [Background] Smith FO, Downey SG, Klapper JA, Yang JC, Sherry RM, Royal RE, Kammula US, Hughes MS, Restifo NP, Levy CL, White DE, Steinberg SM, Rosenberg SA. Treatment of metastatic melanoma using interleukin-2 alone or in conjunction with vaccines. Clin Cancer Res. 2008 Sep 1;14(17):5610-8. doi: 10.1158/1078-0432.CCR-08-0116. PMID 18765555
- [Background] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohorts 1 and 2 did not enroll participants because the study was terminated due to poor accrual.
Groups:
- Cohort 0: Drosophila generated CTL + SQ IL-2
  1 fludarabine, cyclophosphamide, Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ PBL (CTL-05), aldesleukin : Fludarabine 25 mg/m2 x 5 days Cyclophosphamide 60 mg/kg IV x2 days, Up to 1x10e10 CTL-05 cells Aldesleukin 125,000 IU/kg/dose as a daily subcutaneous injection
- Cohort 1: 2 Experimental Lymphodepleting regimen +Cells+Low dose IL-2
  2 fludarabine, cyclophosphamide, Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ PBL, aldesleukin : Fludarabine 25 mg/m2 x 5 days Cyclophosphamide 60 mg/kg IV x2 days, Up to 1x10e10 CTL-05 cells Aldesleukin 125,000 IU/kg/dose as a daily subcutaneous injection
- Cohort 2: 1 Experimental Lymphodepleting regimen +Cells
  3 fludarabine, cyclophosphamide, Drosophila-peptide pulsed Melanoma-reactive autologous CD8+ PBL : Fludarabine 25 mg/m2 x 5 days Cyclophosphamide 60 mg/kg IV x2 days, Up to 1x10e10 CTL-05 cells
Period: Overall Study
Arm/Group | Cohort 0 | Cohort 1 | Cohort 2
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 0 | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 3 |  |  | 3
  >=65 years | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (7.2) |  |  | 53.0 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 2 |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 3 |  |  | 3
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 3 |  |  | 3
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response (CR) is a disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progression disease (PD) is at least a 20 % increase in the sum of the LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 7 months
Population: Cohorts 1 and 2 did not enroll participants because the study was terminated due to poor accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 0 | 0
Participants
  Complete Response | 0 |  |
  Partial Response | 1 |  |
  Progressive Disease | 2 |  |
  Stable Disease | 0 |  |

2. Primary Outcome: Safety of Drosophila Generated PBL Administered in Combination With a Lymphodepleting Preparative Regimen and Supportive Systemic Aldesleukin
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 7 months
Population: Cohorts 1 and 2 did not enroll participants because the study was terminated due to poor accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 0 | 0
Participants | 3 |  |

3. Secondary Outcome: Investigate Low-dose Systemic Aldesleukin to Cell Efficacy
Description: Low-dose systemic aldesleukin will be evaluated to determine cell activity in metastatic melanoma.
Time Frame: 7 months
Population: Zero participants were analyzed for this outcome measure. Greater than 10 participants were needed to evaluate this outcome measure. These were not explored in the small number of patients studied.
Arm/Group | Cohort 0 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Cohort 0 | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 0 (N=3) | Cohort 1 (N=0) | Cohort 2 (N=0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (13) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with unknown ANC <1.0x10e9/L, fever >=3 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No